CLINICAL TRIAL: NCT06365645
Title: Examining the Feasibility and Acceptability of a Novel App-based Cognitive Behavioral Therapy Intervention for Preventing Postpartum Depression
Brief Title: Feasibility & Acceptability of App-based Cognitive Behavioral Therapy for Postpartum Depression Prevention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Adam Lewkowitz, Assistant Professor, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2138752
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Postpartum Depression; Postpartum Anxiety; Stress
Keywords: perinatal mental health; digital health; postpartum depression; postpartum anxiety; smartphone application (app)
MeSH Terms: conditions — Depression, Postpartum; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants who consent will be unaware of the existence of another version of M.Bapp. Obstetric care providers will be aware of participant's enrollment in this trial but not of the study group and will be encouraged to provide standardized care. The research team and outcomes assessors will be blindd to the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- App-based digital parenting education (Active Comparator): App-based digital parenting education will be delivered through a smartphone app with similar features as M.Bapp, but the content delivered through this attention-matched control app will not contain any CBT modules or psychoeducation.
  Interventions: Behavioral: App-based parenting education
- M.Bapp (Experimental): M.Bapp contains the same app-based digital parenting education provided to the active comparator group as well as 9 additional interactive modules based on the MB cognitive behavioral therapy curriculum. M.Bapp contains interactive features and EMA-based voluntary daily assignments that provide the opportunity to receive additional final reimbursement. Those who complete all modules will receive a digital certificate of completion.
  Interventions: Behavioral: M.Bapp

INTERVENTIONS:
Behavioral: M.Bapp — Please see experimental group description.
  Arms: M.Bapp
Behavioral: App-based parenting education — Please see active comparator group description.
  Arms: App-based digital parenting education

SUMMARY:
Postpartum depression (PPD) affects up 10-15% of mothers overall, but the rate of PPD can be as high as 25% among mothers with personal or obstetric risk factors. The Mothers & Babies Program (MB) is a cognitive behavioral therapy (CBT)-based program that has been shown to prevent PPD among high-risk mothers without a prior history of depression. MB has been so consistently effective that the United States Preventive Services Task Force recommends this program be given to high-risk pregnant patients. Originally designed to be given in-person and via groups, MB has been adapted to be given in person one-on-one in clinic or at home and via text message. However, MB has yet to be adapted to a smartphone application (app). Via evidence-based qualitative research and end-user centered design, MB has been adapted to a novel app, M.Bapp. This study aims to examine the feasibility and acceptability of M.Bapp as a study intervention for perinatal patients as well as provide preliminary estimates of effect for the intervention.

DETAILED DESCRIPTION:
Overall, 10-15% of women are diagnosed with postpartum depression (PPD). Though the most significant risk factor for PPD is a history of depression or prior PPD, rates of PPD are as high as 25% among women without prior depression or PPD but with personal risk factors such as reporting little social support or food insecurity during pregnancy and structural factors such as being unmarried. There are profound maternal and pediatric consequences of postpartum mental illness: untreated PPD is associated with maternal morbidity9-11 and impaired child cognitive development. As such, the American College of Obstetricians & Gynecologists recommends screening all postpartum women for PPD.

There are, however, several structural barriers to the implementation of this recommendation. First, to be screened for PPD, women must attend postpartum visits, and <60% of women do so. Barriers such as lack of childcare or transportation reduce postpartum visit attendance and disproportionately affect low-income women. Second, pregnancy-related health insurance ends at 60 days postpartum, but PPD can persist for months after delivery, leaving low-income women without subsidized access to screening or treatment. Third, unlike those with known psychiatric illness, many pregnant women without prior mental illness do not receive antenatal mental health screening (unless via universal screening) leading to delayed recognition of and diagnosis of depressive symptoms. Tools to overcome these barriers are sorely needed, particularly for those with the least access who currently fall through the cracks.

Therapy preventing PPD delivered via smartphone applications (apps) may be such a tool. The USPSTF concluded that Cognitive Behavioral Therapy (CBT) - which teaches coping skills to modify maladaptive conditions, behaviors, and physiological responses24, 25 - reduces rates of PPD by 49%. The USPSTF highlighted the Mothers and Babies (MB) CBT program for reducing rates of PPD by 53% among low-income women of color. MB was originally designed as a preventive in-person therapy for low-income English- and Spanish-speaking women without psychiatric illness and contains one parenting education module and multiple CBT modules. MB has started to become a digital health intervention: online MB has been shown to be feasible, and text-message-base MB has been examined in one small study. However, to our knowledge, no studies of app-based MB exist. Online or text-message MB may increase access, but participation with an app would likely be higher for several reasons. Individuals are more likely to have smartphones than internet access: 96% of those aged 18-29 years own smartphones. Additionally, apps provide two advantages compared to other digital health programs: (1) App-based content is accessible without cellular or internet service, (2) Apps serve as just-in-time adaptive interventions,35-37 delivering support tailored to individual behaviors. Thus, app-based MB may decrease PPD while overcoming barriers to care.

Over the last two years, this NIH-funded study has utilized evidence-based user-centered digital intervention design techniques and qualitative research methodology to adapt the MB curriculum into a novel smartphone application, M.Bapp. Similar to MB, M.Bapp contains one parenting education module and multiple CBT-based modules.We now propose a pilot randomized control trial to examine the feasibility, acceptability, and preliminary estimates of effects of the full MB program via M.Bapp (intervention) when compared to app-based digital parenting education (an attention control group). Our long-term goal is to use M.Bapp to prevent PPD among perinatal women at high-risk for the condition due to those with structural or personal risk factors.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking
* maternal age >18 years old
* smartphone ownership
* receiving prenatal care from a resident or nurse-practitioner/midwifery clinic at the Obstetric and Gynecologic Care Center at WIH
* plan to receive postpartum care at the OGCC,
* gestational age ≥32 weeks'.

Exclusion Criteria:

* Active diagnosis or history within five years of depression, anxiety, or other psychiatric condition, as documented in the electronic medical record
* Endorsing active suicidality on intake survey or screening positive on EPDS (≥10) or Patient Health Questionnaire (PHQ)-9 (≥10) or GAD-7 (≥8)
* prisoners
* inability to consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients must be pregnant in order to participate
Enrollment: 90 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Randomization and six months postpartum
  50% of those who are eligible based on prescreening and who are approached to participate consent to participate and 80% of those randomized to M.Bapp view at least 5 of the 10 modules
Acceptability | Six months postpartum
  Scoring at least 80% on two well-validated scales: the System Usability Scale (focusing on perceived usability of technology) and the Client Satisfaction Questionnaire (focusing on satisfaction with mental health therapy). These surveys will also contain questions covering additional themes about participant experience with the study intervention (either M.Bapp or app-based parenting education)-(1) helpfulness; (2) satisfaction; and (3) ease of interface with technical aspects of the program.

SECONDARY OUTCOMES:
Inventory for Depression Scale | Baseline (32-36 weeks' gestation), within one week of delivery, 2 months postpartum, 4 months postpartum, and 6 months postpartum
  30-item Score from 0 to 84. Screen positive: score ≥26 or suicidal ideation
General Anxiety Disorder-7 | Baseline (32-36 weeks' gestation), within one week of delivery, 2 months postpartum, 4 months postpartum, and 6 months postpartum
  7-item self-report on anxiety symptoms
Perceived Stress-Scale 4 | Baseline (32-36 weeks' gestation), 2 months postpartum, and 6 months postpartum
  4-item self-report on stress symptoms
Dyadic Adjustment Scale | Baseline (32-36 weeks' gestation), 2 months postpartum, and 6 months postpartum
  7-item survey measuring relationship satisfaction, decision-making and cohesion
UCLA Loneliness Scale | Baseline (32-36 weeks' gestation), 2 months postpartum, and 6 months postpartum
  20-item survey measuring loneliness
Frequency of Mothers and Babies Skills Use | 6 months postpartum
  10-item survey created by MB to evaluate perceived helpfulness of intervention

OTHER OUTCOMES:
De novo psychiatric diagnosis | Within one week of delivery, 2 months postpartum, 4 months postpartum, and 6 months postpartum
  Initiation of antidepressant or other psychotropic medication during study period
Screening positive on study survey | Within one week of delivery, 2 months postpartum, 4 months postpartum, and 6 months postpartum
  Screening positive for anxiety, depression, or stress

CONTACTS AND LOCATIONS:
Locations (1):
- Women & Infants Hospital of Rhode Island, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Data from this small pilot will not be made available to other researchers